CLINICAL TRIAL: NCT06187272
Title: Effectiveness of Music on the Performance of Graduate Occupational Therapy Students During
Brief Title: Effectiveness of Music Practical Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russell Sage College (Other)
Responsible Party: Principal Investigator, Christine Mulligan, Assistant Professor, Russell Sage College
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RussellSage
Record Dates: First submitted 2023-11-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Test Anxiety; Stress

STUDY DESIGN:
Intervention Model Description: One group was a control, one group received the intervention
Who Masked: Participant
Masking Description: There was no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one with no music (No Intervention): Graduate students with no music
- Group Two with music (Experimental): Graduate students listening to music
  Interventions: Behavioral: Listening to music

INTERVENTIONS:
Behavioral: Listening to music — Students listened to background music during a practical examination of 60 bpm.
  Arms: Group Two with music

SUMMARY:
College student anxiety is rising alarmingly and directly affects academics, occupations, and well-being. Occupational therapy (OT) students encounter a rigorous workload and pressure to become entry-level practitioners. Higher education faculty strive for evidence-based teaching strategies and effective classroom management and are often challenged to promote a positive classroom culture. This quasi-experimental study explored the effect of listening to music during a lab practical examination on the performance of OT graduate students.

DETAILED DESCRIPTION:
Through convenience sampling, 68 graduate students in an occupational therapy program were recruited to participate. The quasi-experimental study was conducted at Russell Sage College, in Troy, New York, with approval from the International Review Board Inclusion criteria were male and female first and second-year students, ages 19-34, enrolled in Functional Anatomy and Kinesiology or Physical Agent Modalities. The data was collected during lab practicals in December 2021 and June 2023. Forty-three students signed consent forms to participate. Students sign up for 20-minute time slots in pairs for the practical exam. Each student randomly selects confidential assessment cards and takes turns independently completing their assignment. Each practical contains a grading rubric, and a score of 80 is required to pass. Students either had one private room when an examiner during the practical, and either it was quiet or low 60 bpm music played in the background. Pre and post-outcome measures evaluated each student's state, trait, test anxiety, blood pressure, and heart rate outside the assessment room. State and trait anxiety was measured using the State-Trait Anxiety Inventory for Adults™ by Charles D. Spielberger and the Test Anxiety Inventory by Charles D. Spielberger & Associates. State-Trait Anxiety is cited in over 20,000 articles and is the primary assessment used most often for individuals susceptible to anxiety. The reliability of the State-Trait Anxiety is .86 - .95, and substantial evidence confirms its validity. Mean S-anxiety .59, T- T-anxiety .57 college students of both sexes. The Test Anxiety Inventory measures individual situational anxiety of symptom frequency throughout an exam, like apprehension and nervousness. Remote online survey licenses were purchased to administer the State-Trait Anxiety Adult and Test Anxiety Inventory on each student's laptop. Mind Garden's Transform System collected raw scaled scores. The research team recorded blood pressure and heart rate with the digital Blood Pressure monitor with an upper arm cuff.

ELIGIBILITY:
Inclusion Criteria:

* Graduate occupational therapy students enrolled in Functional Anatomy and Kinesiology or Physical Agent Modalities

Exclusion Criteria:

* Students not registered for Functional Anatomy and Kinesiology or Physical Agent Modalities

Ages: 19 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
State-Trait Inventory | Day 1
  The State-Trait Anxiety Inventory a self-report questionnaire, follows a Likert scale and measures state and trait anxiety with 40 questions and a maximum score of 80
Test Anxiety Inventory | Day 1
  The Test Anxiety Inventory is one of the most frequently used self-reported measures of situational anxiety and symptom frequency throughout an exam, like apprehension and nervousness
Blood pressure | Day 1
  The measurement of a systolic and diastolic ratio
Heart rate | Day 1
  Measuring beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Chris Mulligan, Principal Investigator — Russell Sage College
Locations (1):
- Russell Sage College, Troy, New York, United States

IPD SHARING:
Plan to Share IPD: No
Consent form, study protocol, data analysis